CLINICAL TRIAL: NCT05454566
Title: A Single Dose Escalation Study of Intra-Articular ICM-203 in Subjects With Kellgren-Lawrence Grade 2 or Grade 3 Osteoarthritis of the Knee
Brief Title: A Study Evaluating the Safety, Tolerability, and Activity of ICM-203 in Subjects With Knee Osteoarthritis.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ICM Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICM 20-1003
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis, Knee
Keywords: adeno-associated virus; gene therapy; ICM-203; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: * Group 1: ICM-203 6x10e12 vg
  * Group 2: ICM-203 2x10e13 vg
  * Group 3: ICM-203 6x10e13 vg
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: ICM-203 (Low dose) (Experimental): 3 to 6 subjects will receive a single intra-articular injection of ICM-203 at 6x10e12 vg into the target knee at Day 1
  Interventions: Genetic: ICM-203
- Group 2: ICM-203 (Medium dose) (Experimental): 3 to 6 subjects will receive a single intra-articular injection of ICM-203 at 2x10e13 vg into the target knee at Day 1
  Interventions: Genetic: ICM-203
- Group 3: ICM-203 (High dose) (Experimental): 3 to 6 subjects will receive a single intra-articular injection of ICM-203 at 6x10e13 vg into the target knee at Day 1
  Interventions: Genetic: ICM-203

INTERVENTIONS:
Genetic: ICM-203 — Intra-articular injection

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and activity of ICM-203, a recombinant adeno-associated viral (AAV) vector that expresses a therapeutic gene that promotes cartilage formation, reduces joint inflammation and pain, as well as improves joint physical function, by injecting escalating doses of ICM-203 into the knee of subjects with mild to moderate knee osteoarthritis (OA).

Approximately 6 to 18 subjects will be enrolled into 3 successive dose-escalating groups in a 3+3 study design, whereby 3 study subjects in each group will be dosed sequentially with ICM-203 and 3 additional subjects will be dosed at the same dose level if a dose limiting toxicity (DLT) occurs in any of the first 3 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) of 18.0 to 40.0 kg/m2, inclusive, at the time of screening.
2. Kellgren-Lawrence grade 2 or grade 3 OA of target knee.
3. Target knee pain between 4 and 9, inclusive, on an NRS ranging from 0 (no pain) to 10 (worst pain imaginable), at the time of screening.
4. KOOS function in daily living score >25, a measure of knee function ranging from 0 (extreme problems) to 100 (no problems), at the time of screening .
5. A stable treatment regimen for symptomatic relief of OA, including NSAIDs, for 4 weeks prior to screening.

Exclusion Criteria:

1. History of rheumatoid arthritis, psoriatic arthritis, gout, pseudogout, autoimmune OA, chondrocalcinosis, hemochromatosis, villonodular synovitis, and synovial chondromatosis or other disorder that in the opinion of the Investigator could cause inflammation of the knee.
2. Injection of steroid, hyaluronate or other agent, into the target knee less than 90 days prior to day 1.
3. Major injury to the target knee, such as torn ligament or severe sprain, within 12 months of screening.
4. Disability so severe that the subject cannot comply with the study requirements, including knee symptoms that result in significant difficulty or inability to walk.
5. Surgery on the target knee within 180 days prior to day 1.
6. Total knee arthroplasty or other knee surgery planned in the next 12 months.
7. Active joint infection or other concurrent medical or psychiatric condition that, in the opinion of the Investigator, would make the subject unsuitable for the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAEs) | Up to Week 52
  Incidence and Severity of Treatment-Emergent Adverse Events following administration of study drug
Knee pain | Up to Week 52
  Evaluation of change from baseline in knee pain as measured using a Numerical Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable)
Knee function | Up to Week 52
  Evaluation of change from baseline in knee function as measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS) function in daily living subscale ranging from 0 (extreme problems) to 100 (no problems)
Analgesic use | Up to Week 52
  Evaluation of change from baseline in in use of analgesics, such as acetaminophen and NSAIDs
Magnetic Resonance Imaging Osteoarthritis Knee Score (MOAKS) | Up to Week 52
  Evaluation of change from baseline in MOAKS, focusing on articular cartilage and effusion-synovitis
Joint space width | Up to Week 52
  Evaluation of change from baseline in Joint space width in mm as measured on knee radiograph

SECONDARY OUTCOMES:
Humoral response to AAV5.2 capsid | Up to Week 52
  Evaluation of change from baseline in neutralizing antibody titers against AAV5.2 in serum
Cellular immune response to AAV5.2 capsid | Up to Week 52
  Evaluation of change from baseline in T-cell responses to AAV5.2 capsid
Systemic biodistribution of ICM-203 | Up to Week 52
  Evaluation of presence of ICM-203 in peripheral blood after administration of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Alison Heald, MD, Study Director — ICM Co. Ltd.

IPD SHARING:
Plan to Share IPD: No